CLINICAL TRIAL: NCT04547127
Title: A Multicenter, Randomized, Open-label, Parallel Group Pilot Study to Evaluate Safety and Efficacy of Convalescent Methylene Blue Treated (MBT) Plasma From Donors Recovered From Coronavirus Disease 2019 (COVID-19) With Standard Medical Treatment (SMT) Versus SMT Alone in Subjects With COVID-19 Requiring Admission to the Intensive Care Unit (ICU)
Brief Title: A Study to Evaluate Safety and Efficacy of Convalescent Methylene Blue Treated (MBT) Plasma From Donors Recovered From Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC2003; 2020-001299-14 (EudraCT Number)
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: Coronavirus Disease; Severe acute respiratory syndrome coronavirus 2; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent anti-SARS-CoV-2 MBT Plasma + SMT (Experimental): Participants will receive 2 consecutive transfusions of 200 to 250 milliliters (ml) of ABO-compatible convalescent plasma with each unit of plasma, obtained from the same convalescent donor, which will be administered on Day 1 using standard procedures for administration of fresh frozen plasma. Participants weighing less than 45 kilograms (kg) will receive two transfusions of 10 ml of convalescent plasma per kilogram of body weight with each unit of plasma obtained from the same convalescent donor. Participants will also receive all standard of care interventions while hospitalized, from Day 1 to Day 29.
  Interventions: Biological: Convalescent anti-SARS-CoV-2 MBT Plasma; Drug: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Participants will receive all standard of care interventions required throughout the participant's hospitalization, from Day 1 to Day 29.
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Biological: Convalescent anti-SARS-CoV-2 MBT Plasma — Intravenous infusion.
  Arms: Convalescent anti-SARS-CoV-2 MBT Plasma + SMT
Drug: Standard Medical Treatment — SMT

SUMMARY:
The purpose of the study is to determine if Convalescent anti-severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Methylene Blue Treated (MBT) plasma plus Standard Medical Treatment (SMT) can reduce all-cause mortality versus SMT alone in hospitalized participants with COVID-19 requiring admission to the intensive care unit (ICU) through Day 29.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male or female subjects of ≥ 18 years of age at time of Screening who are being treated in the intensive care unit (ICU) for COVID-19 for not longer than 48 hours or for whom a decision has been made that COVID-19 disease severity warrants ICU admission.
* Subject (or a legal representative or a nearest relative or a relative by marriage, as appropriate) provides informed consent (ICF) prior to initiation of any study procedures.
* Has laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by qualitative Polymerase Chain Reaction (PCR) (reverse transcriptase [RT]-PCR), or other commercial or public health assay in any specimen during the current hospital admission prior to randomization.
* Illness (symptoms) of any duration, and the following:

  1. Radiographic infiltrates by imaging (chest x-ray, computerized tomography [CT] scan, etc.), and
  2. Requiring mechanical ventilation and/or supplemental oxygen
* Subjects with no limitation of therapeutic effort (decision on the status and future of the subject).
* Female subjects of child-bearing potential must have a negative test for pregnancy blood or urine human chorionic gonadotropin (HCG)-based assay at Screening/Baseline Visit.

Exclusion Criteria:

* Clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may place the subject at undue medical risk.
* The subject has had a known serious anaphylactic reaction to blood, any blood-derived or plasma product or methylene blue.
* A medical condition in which the infusion of additional fluid is contraindicated.
* Shock unresponsive to fluid challenge and/or multiple vasopressors and accompanied by multiorgan failure considered by the Principal Investigator not able to be reversed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality Rate | Up to Day 29

SECONDARY OUTCOMES:
Change from Baseline in National Early Warning Score (NEWS) | Day 1 through Day 29
Time to Clinical Response as Assessed by NEWS ≤ 2 Maintained for 24 hours | Day 1 through Day 29
Time to Hospital Discharge | Day 1 through Day 29
Time to ICU Discharge | Day 1 through Day 29
Duration of All Oxygen Use | Day 1 through Day 29
Duration of Mechanical Ventilation | Day 1 through Day 29
Absolute Value Change from Baseline in Ordinal Scale | Day 1 through Day 29
Mean Change from Baseline in Ordinal Scale | Day 1 through Day 29
Percentage of Participants in Each Severity Category of the 7-Point Ordinal Scale | Day 15 and Day 29

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Fundación Jimenez Diaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Complejo Hospitalario Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clínico Universitario de Santiago -CHUS, Santiago
  - Hospital Universitari Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No